CLINICAL TRIAL: NCT04643678
Title: Efficacy of Anakinra in the Management of Patients With COVID-19 Infection in Qatar: A Randomized Clinical Trial
Brief Title: Anakinra in the Management of COVID-19 Infection
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Hamad Medical Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MRC-05-140
Record Dates: First submitted 2020-11-24; First posted 2020-11-25 (Actual); Last update posted 2022-08-16 (Actual); Status verified 2021-02

CONDITIONS: Covid19; Pneumonia; Cytokine Release Syndrome; Corona Virus Infection; Viral Infection
MeSH Terms: conditions — COVID-19; Pneumonia; Cytokine Release Syndrome; Coronavirus Infections; Virus Diseases | interventions — Interleukin 1 Receptor Antagonist Protein; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Anakinra Group (Active Comparator): Anakinra + Standard of Care
  Interventions: Drug: Anakinra
- Standard of Care Group (Other): Standard of Care Alone
  Interventions: Other: Standard of Care

INTERVENTIONS:
Drug: Anakinra — Patient will receive Anakinra 100 mg SC injection every 12 hours for 3 days, then 100 mg once daily from day 4 to day 7 plus Standard of Care
  Other Names: Kineret®
  Arms: Anakinra Group
Other: Standard of Care — Patients will receive the Standard of Care therapy as per the local treatment protocol
  Arms: Standard of Care Group

SUMMARY:
Coronavirus Disease 2019 (COVID-19) was first isolated in Wuhan, China in December 2019. It is rapidly spreading worldwide, posing a severe threat to global health. Many therapeutics have been investigated for the treatment of this disease with inconclusive outcomes.

Anakinra - an interleukin (IL)-1 receptor antagonist - had showed survival benefits in patients with macrophage activation syndrome (MAS) and sepsis and was investigated for the use in COVID-19 infection with promising outcomes.

ELIGIBILITY:
Inclusion criteria:

* Hospitalized adult (age ≥ 18yrs)
* Confirmed COVID-19 diagnosis
* Presence of respiratory distress in addition to signs of cytokine release syndrome
* Radiological evidence of pneumonia
* Signed informed consent

Exclusion Criteria:

* Known allergic reactions to the study medication or any component of the product.
* Active bacterial, viral, TB, fungal infectious diseases
* Received immunosuppressant or immunomodulatory in the past 30 days
* Neutrophil count < 500 cells/microliter
* Platelets < 50,000/microliter
* Pregnant or breastfeeding females

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2020-10-30 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Treatment Success at day 14 | Day 14
  Defined as WHO Clinical Progression score of ≤3 [Ambulatory mild disease: symptomatic; assistance needed].

SECONDARY OUTCOMES:
Change in WHO Clinical Progression Score | Day 7
  Change in WHO Clinical Progression Score between day 1 and day 7 [WHO Clinical Progression score: 0 (Uninfected) - 10 (Dead)]
Time to ICU admission | Day 28
  Time to ICU admission up to 28 days
Incidence of Adverse Events | Day 28
  Incidence of adverse events up to 28 days
Length of hospital stay | Day 28
  Length of hospital stay up to 28 days
All-cause Mortality | Day 28
  All-cause mortality rate at hospital discharge or at 28 days, whichever is first

CONTACTS AND LOCATIONS:
Locations (1):
- Hamad Medical Corporation, Doha, Qatar

REFERENCES:
- [Derived] Elmekaty EZI, Maklad A, Abouelhassan R, Munir W, Ibrahim MIM, Nair A, Alibrahim R, Iqbal F, Al Bishawi A, Abdelmajid A, Aboukamar M, Hadi HA, Khattab MA, Al Soub H, Al Maslamani M. Evaluation of anakinra in the management of patients with COVID-19 infection: A randomized clinical trial. Front Microbiol. 2023 Jan 26;14:1098703. doi: 10.3389/fmicb.2023.1098703. eCollection 2023. PMID 36778864